CLINICAL TRIAL: NCT03863717
Title: Investigation of the Effectiveness of Upper Limb Exercise in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University Cyprus (Other)
Collaborators: Nicosia General Hospital (Other)
Responsible Party: Principal Investigator, Christos Karagiannis, PhD candidate in Physiotherapy, European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ΕΕΒΚ/ΕΠ/2017/18
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Endurance Exercise Training Group (Experimental): Pulmonary Rehabilitation Program including Upper Limb Endurance Exercise Training with arm cycle ergometer
  Interventions: Other: Arm Endurance Exercise Training
- Control Group (Active Comparator): Pulmonary Rehabilitation Program without Upper Limb Endurance Exercise Training
  Interventions: Other: Control

INTERVENTIONS:
Other: Arm Endurance Exercise Training — Pulmonary Rehabilitation Program including Upper Limb Endurance Exercise Training with arm cycle ergometer
  Other Names: Pulmonary Rehabilitation
  Arms: Arm Endurance Exercise Training Group
Other: Control — Pulmonary Rehabilitation Program without Upper Limb Endurance Exercise Training
  Other Names: Pulmonary Rehabilitation
  Arms: Control Group

SUMMARY:
The aim of the study is to investigate the efficacy of upper limb exercise training in Chronic Obstructive Pulmonary Disease (COPD) patients. For the purpose of the study, a controlled trial will be conducted within Respiratory Clinic of Nicosia General Hospital. The sample will be divided in two groups. The intervention group will participate in a pulmonary rehabilitation program which includes upper and lower extremities exercises, with addition of arm ergometer. The second group (control group) will participate in the same program but without arm ergometer training.

The study's hypothesis is that the intervention group will improve the outcome measures significantly better than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD confirmed by clinical examination and a pulmonary function test
* Stable clinical condition (without recent respiratory system infections or any exacerbation of the disease)
* Patients must be willing to re evaluate at the end of the study
* Patients must be willing to give written consent for their participation in the study

Exclusion Criteria:

* Age < 18 years old
* Unstable cardiac disease
* Musculoskeletal and neurological diseases that could affect exercise performance or preclude exercise
* Patients of COPD final stage or other serious disease final stage
* Significant cognitive or psychiatric impairment that would lead to an inability to follow simple commands in a group setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Muscle Strength, biceps brachii | Before Intervention
  Assess biceps brachii via hand-held dynamometer Micro FET2
Upper Limb Muscle Strength, biceps brachii | At 3 months (at the end of intervention)
  Assess biceps brachii via hand-held dynamometer Micro FET2
Upper Limb Muscle Strength, biceps brachii | Change from Baseline Biceps Brachii Muscle Strength at 3 months
  Assess biceps brachii via hand-held dynamometer Micro FET2
Upper Limb Muscle Strength, triceps | Before Intervention
  Assess triceps via hand-held dynamometer Micro FET2
Upper Limb Muscle Strength, triceps | At 3 months (at the end of intervention)
  Assess triceps via hand-held dynamometer Micro FET2
Upper Limb Muscle Strength, triceps | Change from Baseline Triceps Muscle Strength at 3 months
  Assess triceps via hand-held dynamometer Micro FET2
Upper Limb Muscle Strength, hand-grip | Before Intervention
  Assess via jamar hand dynamometer
Upper Limb Muscle Strength, hand-grip | At 3 months (at the end of intervention)
  Assess via jamar hand dynamometer
Upper Limb Muscle Strength, hand-grip | Change from Baseline Handgrip Muscle Strength at 3 months
  Assess via jamar hand dynamometer
Dyspnea, modified Borg Scale | Before Intervention
  Assess via modified Borg Scale 0 - 10, 0 = no dyspnea, 10 = maximal dyspnea
Dyspnea, modified Borg Scale | At 3 months (at the end of intervention)
  Assess via modified Borg Scale 0 - 10, 0 = no dyspnea, 10 = maximal dyspnea
Dyspnea, modified Borg Scale | Change from Baseline Dyspnea at 3 months
  Assess via modified Borg Scale 0 - 10, 0 = no dyspnea, 10 = maximal dyspnea
Dyspnea, mMRC Scale | Before Intervention
  Assess via modified Medical Research Council Dyspnea Scale 0 - 4, 0 = breathless only with strenuous exercise, 4 = too breathless to leave the house or breathless when dressing
Dyspnea, mMRC Scale | At 3 months (at the end of intervention)
  Assess via modified Medical Research Council Dyspnea Scale 0 - 4, 0 = breathless only with strenuous exercise, 4 = too breathless to leave the house or breathless when dressing
Dyspnea, mMRC Scale | Change from Baseline Dyspnea at 3 months
  Assess via modified Medical Research Council Dyspnea Scale 0 - 4, 0 = breathless only with strenuous exercise, 4 = too breathless to leave the house or breathless when dressing
Fatigue | Before Intervention
  Assess via modified Borg Scale (0 - 10), 0 = no fatigue, 10 = maximal fatigue
Fatigue | At 3 months (at the end of intervention)
  Assess via modified Borg Scale (0 - 10), 0 = no fatigue, 10 = maximal fatigue
Fatigue | Change from Baseline Fatigue at 3 months
  Assess via modified Borg Scale (0 - 10), 0 = no fatigue, 10 = maximal fatigue
Health-related Quality of Life, SGRQ | Before Intervention
  Assess via Saint George Respiratory Questionnaire, A total score incorporates scores from each component of the SGRQ which ranges from 1 to 100, where 0 indicates best health and 100 indicates worst health
Health-related Quality of Life, SGRQ | At 3 months (at the end of intervention)
  Assess via Saint George Respiratory Questionnaire, A total score incorporates scores from each component of the SGRQ which ranges from 1 to 100, where 0 indicates best health and 100 indicates worst health
Health-related Quality of Life, SGRQ | Change from Baseline at 3 months
  Assess via Saint George Respiratory Questionnaire, A total score incorporates scores from each component of the SGRQ which ranges from 1 to 100, where 0 indicates best health and 100 indicates worst health
Health-related Quality of Life, CAT | Before Intervention
  Assess via COPD Assessment Test (CAT), Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Health-related Quality of Life, CAT | At 3 months (at the end of intervention)
  Assess via COPD Assessment Test (CAT), Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Health-related Quality of Life, CAT | Change from Baseline at 3 months
  Assess via COPD Assessment Test (CAT), Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Activities of Daily Living with Upper Limbs | Before Intervention
  Assess via total time need to perform 3 daily activities: (i) simulating of window cleaning, (ii) dry 10 dishes and putting them on a shelf above shoulder level and (iii) putting three packages, each weighing 1000 g, on a shelf above shoulder level
Activities of Daily Living with Upper Limbs | At 3 months (at the end of intervention)
  Assess via total time need to perform 3 daily activities: (i) simulating of window cleaning, (ii) dry 10 dishes and putting them on a shelf above shoulder level and (iii) putting three packages, each weighing 1000 g, on a shelf above shoulder level
Activities of Daily Living with Upper Limbs | Change from Baseline time at 3 months
  Assess via total time need to perform 3 daily activities: (i) simulating of window cleaning, (ii) dry 10 dishes and putting them on a shelf above shoulder level and (iii) putting three packages, each weighing 1000 g, on a shelf above shoulder level

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, Nicosia General Hospital, Nicosia, Cyprus

REFERENCES:
- [Derived] Karagiannis C, Savva C, Korakakis V, Adamide T, Georgiou A, Matheou I, Prodromou A, Xanthos T. Effect of Strength Versus Strength and Endurance Upper Limb Exercise Training in Patients With Chronic Obstructive Pulmonary Disease: A RANDOMIZED CLINICAL TRIAL. J Cardiopulm Rehabil Prev. 2021 Nov 1;41(6):426-431. doi: 10.1097/HCR.0000000000000620. PMID 34117184